CLINICAL TRIAL: NCT02727621
Title: Dexmedetomidine Based Versus Propofol Based Anesthesia in Patients Undergoing Coronary Revascularization: a Randomized, Double-blind Controlled Study
Brief Title: Dexmedetomidine Sedation and Cardiopulmonary Bypass
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate Professor (Anesthesiology and Critical Care)- College of Medicine-Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB000087801
Record Dates: First submitted 2016-03-30; First posted 2016-04-04 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Coronary Artery Bypass Grafting
Keywords: Dexmedetomidine; Cardiac; Coronary Artery Bypass Grapht; Sedation; Propofol; Intravenous Anesthetics
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine group (Active Comparator)
  Interventions: Drug: Dexmedetomidine
- Propofol group (Active Comparator)
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: Dexmedetomidine — Anesthesia will be maintained with continuous infusion of dexmedetomidine 0.5-0.7 µg/kg/h in addition to sevoflurane supplementation as required, to maintain arterial blood pressure and heart rate within 20% of preoperative values. Muscle relaxation will be maintained with continuous rocuronium infusion 0.6 mg/kg/h.
  Other Names: precedex
  Arms: Dexmedetomidine group
Drug: propofol — Anesthesia will be maintained with continuous infusion of propofol 50-100 µg/kg/min in addition to sevoflurane supplementation as required, to maintain arterial blood pressure and heart rate within 20% of preoperative values. Muscle relaxation will be maintained with continuous rocuronium infusion 0.6 mg/kg/h.
  Other Names: diprivan
  Arms: Propofol group

SUMMARY:
Dexmedetomidine is a unique sedative anesthetic agent that allows accurate control of the depth of sedation and provides analgesia, cardio protection, renal protection, and neuroprotection without causing respiratory depression. It is an alpha 2-adrenoreceptor agonist that modulates the release of catecholamines from the central and autonomic nervous systems. When patients sedated by dexmedetomidine are allowed to become responsive, they are calm and cooperative (1). No other sedative agent has this feature, and sedated patients frequently awaken in a confused state. Investigators are conducting this study project to compare between dexmedetomidine based and propofol based anesthetic techniques with regard to hemodynamic changes, stress hormone release as well as cytokines in patients undergoing CPB for coronary revascularization.

DETAILED DESCRIPTION:
100 patients undergoing elective CPB for coronary revascularization surgery. On the morning of operation the patients were randomized to receive one of two anesthetic techniques dependent on the type of sedation used. Standard anesthetic technique will be used for all patients except for using dexmedetomidine sedation in one group and propofol sedation in the other group.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective coronary revascularization surgery with cardiopulmonary bypass

Exclusion Criteria:

* Severely impaired left ventricular function (ejection fraction <40%)
* Valvular heart disease
* Low cardiac output syndrome
* Uncontrolled rapid atrial fibrillation
* On plavix less than one week
* Severe systemic non-cardiac disease
* Infectious disease
* Poorly controlled diabetes mellitus
* patients on corticosteroids or other immunosuppressive treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
cardiac index | within intraoperative period
  cardiac index measured in L/min/m2

SECONDARY OUTCOMES:
heart rate | within intraoperative period
  heart rate measured in beat/min.
mean arterial blood pressure | within intraoperative period
  mean arterial blood pressure measured in mm.Hg
central venous pressure | within intraoperative period
  central venous pressure measured in mm.Hg
pulmonary capillary wedge pressure | within intraoperative period
  pulmonary capillary wedge pressure measured in mm.Hg
mean pulmonary artery pressure | within intraoperative period
  mean pulmonary artery pressure measure in mm.Hg
systemic vascular resistance index | within intraoperative period
  systemic vascular resistance index measured in dyn.sec/cm5/m2
pulmonary vascular resistance index | within intraoperative period
  pulmonary vascular resistance index measured in dyn.sec/cm5/m2
stroke volume index | within intraoperative period
  stroke volume index measured in ml/m2/beat
left ventricular stroke work index | within intraoperative period
  left ventricular stroke work index measured in gm/m2/beat
cardiac output | within intraoperative period
  cardiac output measured in L/min
inotrope score | 1st 24 hours
  appropriate score
duration of mechanical ventilation | 1st week
  duration of mechanical ventilation measured in hours
sedation score | 1st 24 hours
  appropriate score

CONTACTS AND LOCATIONS:
Overall Officials: Sayed Abd-Elshafy, MD, Principal Investigator — Associate professor, anesthesia and critical care
Locations (1):
- Faculty of Medicine, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided